CLINICAL TRIAL: NCT01508208
Title: A Comparison of Spot Test (Urine Protein/Creatinine Ratio) With 24 - Hour Urine Protein Excretion in Woman With Hypertensive Disorders of Pregnancy
Brief Title: Comparison of Urine Protein/Creatinine Ratio With 24-hour Urine Protein Excretion in Woman With Hypertensive Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research & Development, Saint Thomas Hospital, Panama
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MHST2011-07
Record Dates: First submitted 2012-01-08; First posted 2012-01-11 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2018-01

CONDITIONS: Hypertension, Pregnancy-Induced
Keywords: Hypertension; 24 hour urine protein; Protein/creatinine ratio
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypertensive disorder of pregnancy (Other): Patients with an hypertensive disorder of pregnancy (28 weeks or more of gestation)will collect a random sample of urine for a spot test (protein/creatinine ratio) and urine for 24 hours. The level of proteinuria will be determined in this sample.
  Interventions: Other: Hypertensive disorder of pregnancy

INTERVENTIONS:
Other: Hypertensive disorder of pregnancy — Collection of a random sample of urine for a spot test and a 24 hour urine collection for a 24 hour urine protein.

SUMMARY:
The presence of proteinuria (>300 mg/d) represents an important factor in the diagnosis and evaluation of the pregnant patient with an hypertensive disorder. The 24 hour collection of urine for proteinuria is the gold standard for the diagnosis of the condition and allows the physician to determine if an hypertensive disorder is related directly or not to the gestation.

The problem is the time it takes and the technical difficulties related to the sample collection. An alternative is the quantification of protein and creatinine in a random sample of urine. We seek to evaluate if this method is as affective as the gold standard in the diagnosis of proteinuria (>300 mg/d).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with 28 weeks or more of gestation.
* Complete collection of the 24 hour urine sample.

Exclusion Criteria:

* Failure to recollect the 24 hour urine sample.
* Pregestational Diabetes
* Kidney disease
* 24 hour urine protein > 8.0 g/dL or seric creatinine > 2.0 mg/dL (it could indicate kidney disease).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2012-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity | Six months
  The number of patients with a 24 hour urine collection with a proteinuria > 300mg will be compared with the number of patients with a Spot Test (protein/creatinine ratio in a random urine sample) > 0.2 (equivalent to the 24 hour test > 300 mg). This value will be used to calculate the Sensitivity and Specificity of the spot test.

SECONDARY OUTCOMES:
Positive and Negative Predictive Value | six months
  The number of patients with a 24 hour urine collection with a proteinuria > 300mg will be compared with the number of patients with a Spot Test (protein/creatinine ratio in a random urine sample) > 0.2 (equivalent to the 24 hour test > 300 mg). This value will be used to calculate the positive and negative predective value of the spot test.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo A Reyes, MD, Principal Investigator — Saint Thomas Hospital, Panama; Joanna Buitrago, MD, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas H, Panama City, Panama